CLINICAL TRIAL: NCT05861648
Title: Effect of Folic Acid Supplementation in Patient's Calcific Aortic Valve Disease With Mild Aortic Valve Stenosis
Brief Title: Folic Acid Supplementation in Calcific Aortic Valve Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WUHFACAVD01
Record Dates: First submitted 2023-05-04; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-04

CONDITIONS: Calcification of Aortic Valve; Aortic Valve Stenosis
Keywords: Folic Acid; Calcification of Aortic Valve; Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve, Calcification of; Aortic Valve Stenosis | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Drug group 1 (Experimental): Dietary Supplement: Folic acid 2.5 mg/day
  Interventions: Drug: Folic Acid Oral Tablet
- Control group 2 (Placebo Comparator): Dietary Supplement: Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Folic Acid Oral Tablet — Dietary Supplement: Folic acid 2.5mg/day
  Arms: Drug group 1
Dietary Supplement: Placebo — Dietary Supplement: Placebo
  Arms: Control group 2

SUMMARY:
This is a prospective, randomized, comparative, clinical trial conducted by Wuhan Union Hospital that aims to evaluate the efficacy and safety of folic acid compared to placebo in patients with calcific aortic valve disease with mild aortic valve stenosis.

DETAILED DESCRIPTION:
Folic acid is involved in important physiological activities in the body such as DNA synthesis, cell division and growth and development. Recent studies have shown that folic acid may also have a positive effect on cardiovascular system health. Aortic valve calcification is a cardiovascular disease whose incidence increases progressively with age. Early studies suggest that folic acid may slow the progression of aortic valve calcification by inhibiting cell calcification and promoting calcium deposition. Participants were randomized into two groups: one group was given oral folic acid treatment and the other group was given placebo control. Patients in both groups were observed for aortic valve calcification during the follow-up period, and changes in aortic valve thickness, degree of calcification, and flow were recorded by cardiac ultrasonography, while the incidence of cardiovascular events and adverse effects were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult ≥ 35 years of age at the time of recruiting.
* Subject has calcific aortic valve disease with mild to moderate aortic valve stenosis as defined by Doppler echocardiography results: Aortic Valve mean pressure gradient between 10-30 mmHg and Aortic Valve Area ≥ 1.2 and ≤ 2.0 cm2 on transthoracic echocardiography within 2 weeks prior to randomization and Cardiac Compute Tomography (CT) test results: aortic valve calcium score (Agatston score) ≥ 200 AU at baseline cardiac CT within 1 month prior to randomization
* Subject provides written informed consent prior to initiation of any study procedures.
* Subject understands and agrees to comply with planned study procedures.

Exclusion Criteria:

* Subject has concomitant moderate or severe mitral or tricuspid valve disease.
* Subject has left ventricular ejection fraction < 50%.
* Subject previous history of aortic valve surgery, pancreatitis, malignant tumor, drug or alcohol abuse.
* Subjects whose alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 2.5 times the upper limit of normal range.
* Subjects who cannot undergo Cardiac CT.
* Pregnant or lactating women.
* Consideration by the investigator, for safety reasons, that the subject is an unsuitable candidate to receive study treatment.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Aortic valve calcification | 104 weeks
  Aortic valve calcification as measured by change from baseline in Agatston arbitrary unit (AU) using cardiac computed tomography (CT) at 104 weeks
overall survival | 3 years
  overall survival (OS)

SECONDARY OUTCOMES:
Time-to-major adverse cardiovascular events | 104 weeks
  Time-to-major adverse cardiovascular events of cardiac death, non- fatal myocardial infarction, heart failure hospitalization and stroke
Aortic valve calcification | at week 52
  Change in aortic valve calcification as measured by Agatston AU using cardiac computed tomography (CT) at week 52
Change in aortic valve stenosis severity | at week 104
  Change in aortic valve stenosis severity as measured by peak transaortic velocity using echocardiography at week 104 as compared to baseline

IPD SHARING:
Plan to Share IPD: Yes
we would like to share individual participant data with other researchers 1 years after the trial completely finished
Supporting Information: Study Protocol, ICF, CSR
Access Criteria: All data should only be used for academic research.

REFERENCES:
- [Background] Gao L, Chalupsky K, Stefani E, Cai H. Mechanistic insights into folic acid-dependent vascular protection: dihydrofolate reductase (DHFR)-mediated reduction in oxidant stress in endothelial cells and angiotensin II-infused mice: a novel HPLC-based fluorescent assay for DHFR activity. J Mol Cell Cardiol. 2009 Dec;47(6):752-60. doi: 10.1016/j.yjmcc.2009.07.025. Epub 2009 Aug 3. PMID 19660467
- [Background] Moens AL, Claeys MJ, Wuyts FL, Goovaerts I, Van Hertbruggen E, Wendelen LC, Van Hoof VO, Vrints CJ. Effect of folic acid on endothelial function following acute myocardial infarction. Am J Cardiol. 2007 Feb 15;99(4):476-81. doi: 10.1016/j.amjcard.2006.08.057. Epub 2006 Dec 28. PMID 17293188
- [Background] Shirodaria C, Antoniades C, Lee J, Jackson CE, Robson MD, Francis JM, Moat SJ, Ratnatunga C, Pillai R, Refsum H, Neubauer S, Channon KM. Global improvement of vascular function and redox state with low-dose folic acid: implications for folate therapy in patients with coronary artery disease. Circulation. 2007 May 1;115(17):2262-70. doi: 10.1161/CIRCULATIONAHA.106.679084. Epub 2007 Apr 9. PMID 17420345
- [Background] Stanger O. Physiology of folic acid in health and disease. Curr Drug Metab. 2002 Apr;3(2):211-23. doi: 10.2174/1389200024605163. PMID 12003352
- [Background] Gao L, Siu KL, Chalupsky K, Nguyen A, Chen P, Weintraub NL, Galis Z, Cai H. Role of uncoupled endothelial nitric oxide synthase in abdominal aortic aneurysm formation: treatment with folic acid. Hypertension. 2012 Jan;59(1):158-66. doi: 10.1161/HYPERTENSIONAHA.111.181644. Epub 2011 Nov 14. PMID 22083158